CLINICAL TRIAL: NCT03845374
Title: Prospective, Randomized Multi-Center Study of Using the Hyper-CL™ Lens in Subjects Suffering From Bacterial Keratitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye-yon Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLI-H004
Record Dates: First submitted 2019-02-07; First posted 2019-02-19 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Bacterial Keratitis

STUDY DESIGN:
Intervention Model Description: 40 patients will be randomized to one of the following 2 groups:
  * Treatment Group 1: Conventional treatment of topical Antibiotics+ Hyper-CL lens
  * Treatment Group 2: Conventional treatment with topical Antibiotics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Antibiotics+ Hyper-CL™ lens (Experimental): Conventional treatment with topical Antibiotics+ Hyper-CL™ lens
  Interventions: Device: Hyper-CL™ lens
- Conventional Antibiotics (No Intervention): Conventional treatment with topical Antibiotics

INTERVENTIONS:
Device: Hyper-CL™ lens — Use of the Hyper-CL™
  Arms: Conventional Antibiotics+ Hyper-CL™ lens

SUMMARY:
This study is a prospective, randomized, open-label, two arms, clinical study aim to evaluate the efficacy and safety of treatment with Hyper-CL™ lens + Antibiotics compared with treatment with Antibiotics only, in subjects with Bacterial keratitis.

The design of the Hyper-CL™ lens increases contact time of the antibiotics on the cornea enabling increased bioavailability of the active drug.

DETAILED DESCRIPTION:
The Hyper-CL™ Therapeutic soft contact lenses for short-term wear (up to 7 days) are indicated for therapeutic use to promote corneal healing and relieve corneal pain by protecting the cornea during the treatment of acute or chronic pathologies, such as corneal edema, corneal erosions, entropion, bullous keratopathy, and corneal dystrophies as well as post-surgical conditions resulting from cataract extraction and corneal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18-86 years old
2. Subject with Bacterial keratitis in one eye only
3. Subject with Bacterial Keratitis of at least grade 2 score in Average length of infiltration and in Average length of epithelial defect (1mm or above)
4. Best-corrected visual acuity of 6/60 or better in the uninvolved eye
5. No prior antibiotic treatment for current Bacterial Keratitis
6. Subject understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed

Exclusion Criteria:

1. Perforation or imminent perforation of cornea
2. Subject with glaucoma shunts (e.g. Ahmed valve) and or bleb
3. Sign of inflammation in both eyes
4. Severe itching suggesting viral infection or allergy reaction
5. Subepithelial infiltrate suggesting viral infection
6. Dendrite like ulcer or suspecting of Herpes keratitis
7. Previous penetrating keratoplasty
8. No light perception in the affected eye
9. Pregnancy
10. Other active ocular infection
11. Any infiltration suggesting other than bacterial infection e.g. parasite, fungal
12. Any corneal transplant
13. Post refractive surgery
14. Corneal inlays
15. Any other condition which in the opinion of the investigator would place the patient at undue risk for participation.
16. Participation in another clinical study within the past 30 days

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Change in Bacterial Keratitis severity score | From date of randomization up to 14 days
  Will be measured by Bacterial keratitis severity score (0-5). A low score is considered an improvement, a high score is considered worsening.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Rambam Medical Center, Haifa
  - Sheba Medical Center, Ramat Gan